CLINICAL TRIAL: NCT01873053
Title: A 12 Week, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel, Phase II Trial to Evaluate the Efficacy and Safety of WIN-34B in Patients With Osteoarthritis of the Knee
Brief Title: A 12 Week, Phase II Trial to Evaluate the Efficacy and Safety of WIN-34B in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other); Hamsoa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Park Dong-Suk, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KR-KHNMC-OA02
Record Dates: First submitted 2013-05-22; First posted 2013-06-07 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; WIN-34B
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — WIN 34B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1st group : WIN-34B 900mg (Experimental): Patients assigned to 1st group take WIN-34B 450mg BID for 12weeks
  Interventions: Drug: WIN-34B
- 2nd group : WIN-34B 1800mg (Experimental): Patients assigned to 2nd group take WIN-34B 900mg BID for 12weeks
  Interventions: Drug: WIN-34B
- 3rd group : Placebo (Placebo Comparator): Patients assigned to 3rd group take Placebo BID for 12weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WIN-34B — Patients assigned to Experimental group(1st or 2nd group) take WIN-34B 450mg or WIN-34B 900mg BID for 12weeks
  Arms: 1st group : WIN-34B 900mg; 2nd group : WIN-34B 1800mg
Drug: Placebo
  Arms: 3rd group : Placebo

SUMMARY:
This trial is a multi-center, randomized, double-blind, placebo-controlled, parallel, phase II clinical trial and aimed at osteoarthritis of the knee.

Patients who signed informed consent voluntarily and eligible for this study are assigned randomly to one of 3 groups after 2 week-Washout period.

1. st group (experimental) : WIN-34B 450mg BID
2. nd group (experimental) : WIN-34B 900mg BID
3. rd group (Comparator) : Placebo BID

Patients will take WIN-34B or Placebo BID for 12 weeks. Based on baseline, after 4 weeks(Visit 3) and 12 weeks(Visit 5), Researchers check patients' physical examination, questionnaire, laboratory experiment.

After 8 weeks(Visit 4), researchers check adverse effects and current medication status via telephone interview.

After 12 weeks(Visit 5) patients stop taking drugs and after 16 weeks(Visit 6) researchers check patients' physical examination, questionnaire, adverse effects and current medication status.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 35 and 80 years of age
2. Diagnosed with Osteoarthritis of the knee at least 3 months
3. Diagnosed with Osteoarthritis of the knee, based on ACR criteria
4. Able to communicate with researchers and write questionnaires
5. At the screening visit, checking 100mm Pain VAS at least 80mm
6. At randomization(Visit 2), checking 100mm Pain VAS over 50mm
7. Agreeing to participate and signing informed consent voluntarily

Exclusion Criteria:

1. Previous intra-articular injection on knee within 3 months
2. Previous knee surgery within 6 months or scheduled procedures
3. Other diseases that could affect or interfere with the therapeutic outcomes
4. Experiencing habitual use of psychotropic, narcotic analgesic drugs over 1 week
5. Diagnosed with gastrointestinal diseases, unable to stop medicines during the study
6. At the screening visit, identified liver dysfunction
7. At the screening visit, identified renal dysfunction
8. Patients who cannot take NSAIDs
9. Pregnancy and breast-feeding (women of childbearing age need pregnancy test)
10. Physicological or mental disorders, including drug-takers
11. Orthopedic diseases that could affect or interfere with the therapeutic outcomes
12. Inappropriate for the study

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
KWOMAC(Korean Western Ontario and McMaster Universities Osteoarthritis Index) | Changes from baseline at 4, 12, 16weeks

SECONDARY OUTCOMES:
Pain VAS 100mm | Visit1(screening), Visit2(0week), Visit3(4weeks), Visit4(8weeks), Visit5(12weeks), Visit6(16weeks)
KHAQ(Korean Health Assessment Questionnaire) | Visit2(0week), Visit3(4weeks), Visit5(12weeks), Visit6(16weeks)
LFI(Lequesne's Functional Index) | Visit2(0week), Visit3(4weeks), Visit5(12weeks), Visit6(16weeks)
Nine Point Scale | Visit5(12weeks)
Cold-Heat Questionnaire | Visit2(0week), Visit3(4weeks), Visit5(12weeks), Visit6(16weeks)
Dose and Frequency of Rescue drug | Visit2(0week), Visit3(4weeks), Visit4(8weeks), Visit5(12weeks), Visit6(16weeks)
Safety(Vital sign, Physical examination, Laboratory experiment, ECG, Adverse event) | Visit1(screening), Visit2(0week), Visit3(4weeks), Visit4(8weeks), Visit5(12weeks), Visit6(16weeks) - There are some differences in subgroup at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Suk Park, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Oriental Medicine Hospital at Gangdong, Seoul, South Korea